CLINICAL TRIAL: NCT03107572
Title: Comparison of the Predictive and Prognostic Value of Cellular Dysoxia Markers in the Postoperative Period of Cardiac Surgery With Extracorporeal Circulation
Brief Title: Predictive and Prognostic Value of Cellular Dysoxia Markers After Cardiac Surgery With Extracorporeal Circulation
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: NI_2016; IRB 00010254 --2016-030 (Other: IRB number, SFAR); DEC2015-136 (Other: Cnil number by CHRU Lille)
Record Dates: First submitted 2017-03-15; First posted 2017-04-11 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; Microcirculation; Tissue Oxygenation; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples in All patients, Microcirculation reactivity using thenar StO2 and vascular occlusion test, VCO2 and VO2 measurement using indirect calorimetry (at the discretion of attending physician)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study consist of evaluation in cardiac surgery with cardiopulmonary bypass (CPB) setting the ability of PCO2 derived variables (ΔPCO2, ΔPCO2/C(a-v)O2 ratio), compared to lactate and ScVO2 to predict major postoperative adverse events.

DETAILED DESCRIPTION:
Cardiac surgery with cardiopulmonary bypass is associated with serious morbidity and mortality especially in moderate and high-risk patients. This procedure is associated with systemic inflammatory response as a consequence of cardiopulmonary bypass, surgical insult and genetic background of patients leading to organ injury and worse outcome. This pitfall may be worsened by hemodynamic changes with inadequate hemodynamic management.

During and after CPB, substantial changes in macrocirculation and microcirculation are observed and sustain impairment may result in reduced oxygen delivery and/or impaired oxygen extraction. The main consequence is cellular dysorexia that may trigger postoperative organ dysfunction. Rapid identification of cellular dysorexia and rapid hemodynamic management are therefore among key strategies that may reduce mortality.

In this purpose various marker can be considered. Traditionally lactatemia is considered as surrogate of anaerobic metabolism resulting from ischemia. However it interpretation may be challenging particularly in case of reduced hepatic clearance, use of epinephrine or massive blood transfusion. Venous or central venous oxygenation (S(c)VO2), a surrogate of oxygen extraction that is believed to reflect balance between oxygen delivery and consumption, is considered as an acceptable alternative as it was shown to be associated with organ dysfunction in various clinical setting. Nevertheless ScVO2 suffers from the difficulties to define adequate threshold as very high S(c)VO2 as well as low S(c)VO2 may be associated with poor outcome. Recently PCO2 derived dysorexia and perfusion markers have been shown to be predicting outcome in both septic patient and high risk surgical patient. Central venous to arterial difference in PCO2 (ΔPCO2) a global perfusion index is show to be correlated to microcirculation dysfunction and may reflect impaired tissue perfusion. In high risk non-cardiac surgical patients and in septic patient, ΔPCO2 predicted worse outcome better than S(c)VO2 and lactate. Besides this performance may be improve when using a clinically available surrogate based on ΔPCO2. When anaerobic metabolism occurred as a result of sustained hypoxia, CO2 production increases therefore the respiratory quotient (CO2 production (VCO2) and oxygen consumption (VO2) ratio) increases. VCO2/VO2 can be simplified as ΔPCO2 /Ca-vO2 ratio, where Ca-vO2 is arteriovenous O2 content difference. All these variables have never been compared in cardiac surgery setting and their association with microcirculation impaired is poorly documented. The hypotheses is that ΔPCO2, and ΔPCO2 /Ca-vO2 ratio may better predict major postoperative adverse events than blood lactate and S(c)VO2 after cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Cardiac surgery with cardiopulmonary bypass
* Tip of a central venous catheter positioned in superior vena cava or right atria
* Arterial catheter correctly positioned

Exclusion Criteria:

* KDIGO 3 AKI prior to surgery
* Hepatic insufficiency prior to surgery
* Extracorporeal life support prior to surgery '
* Live expectancy lower than 48 hours
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with cardiopulmonary bypass in the university hospital of Lille.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Performances of PCO2 derived perfusion markers (ΔPCO2 and ΔPCO2/C(a-v)O2 ratio) measured 2 hours after CPB to predict major postoperative adverse events (MPAE) in the 48 hours following cardiac surgery. | First 2 days after surgery
  Composite outcome defined as:
  * Acute kidney injury (AKI) with KDIGO score of 2 or more
  * Acute myocardial infarction according to the universal definition of acute myocardial ischemia
  * ARDS according to Berlin definition or respiratory failure (P/F ratio < 300 mmHg + need of mechanical ventilation)
  * Stroke or generalized seizure
  * Cardiogenic or distributive shock defined as hypotension (SAP <90 mmHg, MAP< 65 mmHg) and reduced of cardiac index, ejection fraction or worsening of previously known reduce cardiac index or ejection fraction.
  * Revision surgery
  * Hemorrhagic shock
  * Death

SECONDARY OUTCOMES:
Performances of PCO2 derived perfusion marker measured ICU admission, 6 and 24 hours after CPB to predict major postoperative adverse events (MPAE) in the 2 and 7 days following cardiac surgery. | 2 and 7 days following cardiac surgery
Performances of PCO2 derived perfusion marker measured ICU admission, 6 and 24 hours after CPB to predict organ failure (any organ failure with specific SOFA of 2 or more) in the 2 and 7 days after surgery. | 2 and 7 days following surgery
Kinetics and relation of PCO2 derived variables, lactate and ScVO2 in the 24 hours following surgery. | 24 hours following surgery
Association of CO2 derived variables with lactate clearance, vasopressive score and outcome variables (ICU and hospital length of stay, ICU and hospital mortality). | 24 hours following surgery

OTHER OUTCOMES:
Relation of thenar StO2 with vascular occlusion test derived variables and cellular dysorexia and perfusion markers, and their predictive value in postoperative complication after cardiac surgery. | 2 and 7 days following surgery
Association of PCO2 derived variables, lactate, ScVO2, StO2 derived variables with VO2, VCO2 and respiratory quotient (measured using indirect calorimetry). | 24 hours following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mouhamed MOUSSA, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service d'Anesthésie-Réanimation CCV Hôpital Cardiologique Centre Hospitalier et Universitaire de Lille, Lille, NORD, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shahbazi S, Khademi S, Shafa M, Joybar R, Hadibarhaghtalab M, Sahmeddini MA. Serum Lactate Is not Correlated with Mixed or Central Venous Oxygen Saturation for Detecting Tissue Hypo Perfusion During Coronary Artery Bypass Graft Surgery: A Prospective Observational Study. Int Cardiovasc Res J. 2013 Dec;7(4):130-4. Epub 2013 Dec 1. PMID 24757637
- [Result] Laine GA, Hu BY, Wang S, Thomas Solis R, Reul GJ Jr. Isolated high lactate or low central venous oxygen saturation after cardiac surgery and association with outcome. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1271-6. doi: 10.1053/j.jvca.2013.02.031. Epub 2013 Sep 5. PMID 24011873
- [Result] Balzer F, Sander M, Simon M, Spies C, Habicher M, Treskatsch S, Mezger V, Schirmer U, Heringlake M, Wernecke KD, Grubitzsch H, von Heymann C. High central venous saturation after cardiac surgery is associated with increased organ failure and long-term mortality: an observational cross-sectional study. Crit Care. 2015 Apr 16;19(1):168. doi: 10.1186/s13054-015-0889-6. PMID 25888321
- [Result] Futier E, Robin E, Jabaudon M, Guerin R, Petit A, Bazin JE, Constantin JM, Vallet B. Central venous O(2) saturation and venous-to-arterial CO(2) difference as complementary tools for goal-directed therapy during high-risk surgery. Crit Care. 2010;14(5):R193. doi: 10.1186/cc9310. Epub 2010 Oct 29. PMID 21034476
- [Result] Gasparovic H, Gabelica R, Ostojic Z, Kopjar T, Petricevic M, Ivancan V, Biocina B. Diagnostic accuracy of central venous saturation in estimating mixed venous saturation is proportional to cardiac performance among cardiac surgical patients. J Crit Care. 2014 Oct;29(5):828-34. doi: 10.1016/j.jcrc.2014.04.012. Epub 2014 Apr 26. PMID 24857639
- [Result] Robin E, Futier E, Pires O, Fleyfel M, Tavernier B, Lebuffe G, Vallet B. Central venous-to-arterial carbon dioxide difference as a prognostic tool in high-risk surgical patients. Crit Care. 2015 May 13;19(1):227. doi: 10.1186/s13054-015-0917-6. PMID 25967737
- [Result] Ospina-Tascon GA, Umana M, Bermudez W, Bautista-Rincon DF, Hernandez G, Bruhn A, Granados M, Salazar B, Arango-Davila C, De Backer D. Combination of arterial lactate levels and venous-arterial CO2 to arterial-venous O 2 content difference ratio as markers of resuscitation in patients with septic shock. Intensive Care Med. 2015 May;41(5):796-805. doi: 10.1007/s00134-015-3720-6. Epub 2015 Mar 20. PMID 25792204
- [Result] Mallat J, Lemyze M, Meddour M, Pepy F, Gasan G, Barrailler S, Durville E, Temime J, Vangrunderbeeck N, Tronchon L, Vallet B, Thevenin D. Ratios of central venous-to-arterial carbon dioxide content or tension to arteriovenous oxygen content are better markers of global anaerobic metabolism than lactate in septic shock patients. Ann Intensive Care. 2016 Dec;6(1):10. doi: 10.1186/s13613-016-0110-3. Epub 2016 Feb 3. PMID 26842697
- [Derived] Moussa MD, Durand A, Leroy G, Vincent L, Lamer A, Gantois G, Joulin O, Ait-Ouarab S, Deblauwe D, Caroline B, Decoene C, Vincentelli A, Vallet B, Labreuche J, Kipnis E, Robin E. Central venous-to-arterial PCO2 difference, arteriovenous oxygen content and outcome after adult cardiac surgery with cardiopulmonary bypass: A prospective observational study. Eur J Anaesthesiol. 2019 Apr;36(4):279-289. doi: 10.1097/EJA.0000000000000949. PMID 30664011